CLINICAL TRIAL: NCT06380712
Title: HyperTessa User Experience Study: Evaluation of Acceptance for a Digital Health Solution That Supports the Management of the Hypertensive Condition
Brief Title: HYPERTESSA "HyperTessa User Experience Study (HTUX)"
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Flex Andrea, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6509
Record Dates: First submitted 2024-03-28; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Hypertension
Keywords: Hypertension; Blood pressure; Cardiovascular diseases; Digital health solution
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Hypertension is the primary cause of cardiovascular diseases and premature death in the world. Hypertension management starts with the control of blood pressure, whatever it is the type and severity. The optimum control of blood pressure requires regular and frequent auto-monitoring of blood pressure values, adherence to medication plan, and modification of lifestyle behaviours, including diet, quit smoking, and physical activity. This study is a pilot project to assess acceptance ad usability of a digital health solution to be used by patients diagnosed with hypertension. Materials and methods: Prior to the development of the solution, a literature research was performed, then focus group meetings were conducted with senior experts in the digital field, physicians treating hypertension, and patients. A mobile app and web platform were created to help patients in monitoring and reporting data about health status and lifestyle. In order to execute the study, first the physicians in charge of the study will register in the webApp, creating a personal account. Then, patients who meet the inclusion criteria are proposed to participate to the study and, in case of agreement, will be asked to sign the informed consent (IC) statement and the privacy policy. After the phase of profile setting and onboarding, the patient will start to use the mobile App for hypertension management. Once the patient has used the App for the observation period, the physician will be allowed to analyze the data to understand the level of acceptance and regular usage from each patient. This physician will perform this analysis using a web-based portal which is part of the digital solution. Results: During the study, data about usage patterns will be collected. Specific data about usability and acceptance will be gathered through the use of User Experience Questionnaire (UEQ) and unstructured interviews and tests. After each patient has completed the observation period, all the data will be analysed using mainly descriptive statistics to obtain metrics related to usage patterns, usability and adherence. The study results from this pilot phase will be used to modify the digital solution, leveraging an incremental, iterative logic following a co-design and agile methodology. After incorporating the feedback from this pilot and further enriching the solution, next phases of the study are forseen in order to assess the care benefit of such technology in terms of improved treatment outcomes, due to better adherence, higher motivation in practicing healthy lifestyle, better information, and personalized support from HCP.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years or older;
* Evidence of hypertension, including newly diagnosed, according to the criteria of the European Society of Cardiology (https://www.escardio.org/Guidelines/Clinical-Practice-Guidelines/Arterial-Hypertension-Management-of);
* Patients currently being treated with antihypertensive drugs (regardless of reported blood pressure values): beta blockers, calcium channel blockers, diuretics (any type), alpha-1 lytics, ACE inhibitors, Sartans (at least 1 drug belonging to at least 1 class of that listed);
* Owners of smartphones with compatible operating system;
* To be enrolled in the study and start observation period, patients will first be asked to test the use of the App for fifteen days, verify with him/her any blocking points, validate full comprehension and confirm willingness to participate (run-in phase);
* Subjects must be able to provide written informed consent.

Exclusion Criteria:

* Patients who need to take medication therapy more than twice a day;
* Pregnant patients or women planning to conduct a pregnancy during the course of the study;
* Diagnosis of persistent or permanent atrial fibrillation;
* Subjects with advanced renal failure (eGFR ≤ 15 ml/min/1.73 m2, estimated by MDRD formula) on dialysis treatment (hemodialysis or peritoneal dialysis);
* Subjects with advanced forms of hearing loss such that they are unable to sustain a telephone or face-to-face conversation easily;
* Subjects unable to speak fluently Italian language;
* Patients undergoing chemotherapy and/or radiation treatment or for whom one and both of these treatments are scheduled to begin during the study;
* Diagnosis of terminal cancer (whether or not radio/chemotherapy treatment is present);
* Diagnosis of dementia;
* Diagnosis of psychosis;
* Diagnosis of mental impairment;
* Subjects with heart failure with NYHA functional class III or IV;
* Patients with congenital heart disease, hypertrophic cardiomyopathy and severe aortic stenosis;
* Patients with recent (within 90 days of enrollment date) acute cardio-cerebrovascular event (unstable angina, STEMI and NSTEMI type myocardial infarction, TIA, stroke) and/or with recent (within 90 days of enrollment date) invasive procedure (coronary angioplasty, carotid angioplasty, coronary artery bypass grafting, any other cardiac surgery for which extracorporeal circulation was used);
* Established or suspected forms of secondary hypertension;
* Subjects enrolled in other studies;
* Evidence of severe forms of hypertension, according to the criteria of the European Society of Cardiology (https://www.escardio.org/Guidelines/Clinical-Practice Guidelines/Arterial-Hypertension-Management-of);
* Systolic blood pressure, assessed by noninvasive method (sphingomanometer), ≥ 180 mmHg;
* Diastolic blood pressure, assessed by noninvasive method (sphingomanometer), ≥ 110 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with arterial hypertension aged 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-02 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
User Experience / User Acceptance Indicators for patients | 1 month follow-up
  Acceptance rate above 70% (ratio of patients who were proposed to participate vs patients enrolled); % of patients who don't complete at least 4 assessments in a row (2 weeks usage), max 25%; % of patients who request to dropout the study before the minimum observational period (1 month), max 25%; min 70% of assessments completed by patients; average result of User Experience Questionnaire (UEQ) for all patients: minimum "Good"

SECONDARY OUTCOMES:
User Experience / User Acceptance Indicators for Healthcare Professionals | 1 month follow-up
  • Average result of User Experience Questionnaire (UEQ): minimum "Good"

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Flex, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli., IRCCS, Rome, Italy